CLINICAL TRIAL: NCT00354237
Title: Effect of Strict Glycemic Control on Improvement of Exercise Capacities (VO2 Peak, Peak Workload After Cardiac Rehabilitation, in Patients With Type 2 Diabetes Mellitus With Coronary Artery Disease.
Brief Title: DARE: Diabetes in cArdiac REhabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Principal Investigator, Prof. Bruno Vergès, Professor, Centre Hospitalier Universitaire Dijon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DGS2005/0130
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Type 2 Diabetes Mellitus; Coronary Artery Disease
Keywords: diabetes mellitus; cardiac rehabilitation; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Other): No intensive treatment
  Interventions: Other: Conventional antidiabetic treatment
- A (Experimental): Intensive insulin treatment
  Interventions: Other: Intensive insulin treatment

INTERVENTIONS:
Other: Conventional antidiabetic treatment — No intensive treatment
  Arms: B
Other: Intensive insulin treatment — Intensive insulin treatment
  Arms: A

SUMMARY:
The aim of the DARE study is to see whether strict glycemic control during cardiac rehabilitation may ameliorate the improvement of exercise capacities (VO2 peak, peak workload, ventilatory threshold)in patients with type 2 diabetes with coronary artery disease.

DETAILED DESCRIPTION:
In a recent study, we showed that the benefit of cardiac rehabilitation on the improvement of exercise capacities (VO2 peak, peak workload, ventilatory threshold), after an acute coronary event, was significantly reduced in patients with type 2 diabetes. Moreover ,we showed, in multivariate analysis, that the worse improvement of the capacities to the effort after cardiac rehabilitation, was mainly related to hyperglycemia.

Because the improvement of exercise capacities after cardiac rehabilitation (in particular VO2 peak) has been shown to be an essential factor to reduce short- term and long-term morbidity and mortality, we may think that such benefit on reduction of morbidity and mortality may be significantly less in patients with diabetes.

Thus, we propose to carry out a multicentric intervention study, entitled DARE which goal is to see whether a strict glycemic control, during cardiac rehabilitation following an acute Myocardial Infarction (MI), is likely to improve, the results of cardiac rehabilitation on exercise capacities in patients with type 2 diabetes.

After arrival in cardiac rehabilitation, patients with diabetes, will be randomized into 2 groups: an "intensive treatment" group, in which the patients will treated by insulin under a basal-bolus regimen with strict glycemic control and a "conventional treatment" group, in which the previous anti-diabetic treatment will be continued.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* recent Miocardial Infarction
* HbA1c above 7%
* enrolled in a cardiac rehabilitation program

Exclusion Criteria:

* Type 1 diabetes
* Coronary Bypass Surgery
* Renal Failure (creatinine clearance below 30 ml/min)
* severe Respiratory Failure

Ages: 25 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
improvement of peak VO2, | at the beginning and at the end of the cardiac rehabilitation programm
  Effect of strict glycemic control during cardiac rehabilitation on improvement of peak VO2.For this purpose, we paln to compare first the 2 treatment groups (intensive vs. control) and second, 2 pre-specified glycemic control groups according to the final fructosamine level (below and above the median).

SECONDARY OUTCOMES:
number of patients, in each group of treatment, having improved from at least 16% their peak VO2, after cardiac rehabilitation. | at the beginning and at the end of the cardiac rehabilitation programm
study of the influence of improvement of glycemic control on the results of cardiac rehabilitation on exercise capacities (peak of VO2, peak workload , ventilatory threshold). | at the beginning and at the end of the cardiac rehabilitation programm
improvement of ventilatory threshold | from the beginning and at the end of the cardiac rehabilitation programm
  Effect of strict glycemic control during cardiac rehabilitation on improvement of ventilatory threshold

CONTACTS AND LOCATIONS:
Overall Officials: Bruno L Vergès, Prof, Principal Investigator — Centre Hospitalier Universitaire Dijon
Locations (12):
- France (12):
  - Centre hospitalier du pays d'Aix, Aix-en-Provence
  - Clinique Rhône Durance, Avignon
  - Hôpital J Minjoz, Besançon
  - CMC Bligny, Briis-sous-Forges
  - centre de réadaptation cardiaque "Château le moine", Cenon
  - CHU du Bocage, Dijon
  - Centre IRIS, Marcy-l'Étoile
  - Centre Hospitalier de MONTBARD, Montbard
  - Hopital BROUSSAIS, APHP, Paris
  - Hôpital du haut Lévêque, Pessac
  - Rééducation cardiovasculaire CRF Kerpape, Ploemeur
  - Hôpital jeanne d'arc, Toul

REFERENCES:
- [Derived] Verges B, Patois-Verges B, Iliou MC, Simoneau-Robin I, Bertrand JH, Feige JM, Douard H, Catargi B, Fischbach M; DARE Study group. Influence of glycemic control on gain in VO2 peak, in patients with type 2 diabetes enrolled in cardiac rehabilitation after an acute coronary syndrome. The prospective DARE study. BMC Cardiovasc Disord. 2015 Jul 8;15:64. doi: 10.1186/s12872-015-0055-8. PMID 26152221